CLINICAL TRIAL: NCT04087785
Title: microRNA Profile Associated With Positive Lymph Node Metastasis in Early-stage Cervical Cancer
Brief Title: microRNA Profile in Early-stage Cervical Cancer
Status: Completed | Type: Observational
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, David Cantu, Chief of clinical trials department, National Institute of Cancerología
Other Study IDs: Rev/06/15
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Cervical Cancer
Keywords: miRNAs; cervical cancer; lymph node metastasis
MeSH Terms: conditions — Uterine Cervical Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded tissue blocks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive metastasis: Positive occult lymph node metastasis pathology
- Negative metastasis: Without lymph node metastasis pathology

SUMMARY:
Persistent infections with high-risk subtypes of the human papillomavirus (HPV) are recognized as the etiological factor for developing cervical cancer. The aim od this study was to identify a miRNA profile in patients with early-stage cervical cancer with positive lymph node metastasis treated. Formalin-fixed paraffin-embedded (FFPE) tissue samples of patients with a diagnosis of early-stage cervical cancer treated by radical hysterectomy with lymphadenectomy were collected.

DETAILED DESCRIPTION:
Cervical carcinoma (CC) is one of the most common cancers in women from countries with emerging economies; in Mexico, CC has the second highest incidence and mortality rate. Several studies have demonstrated that the most important prognostic factor is lymph node metastasis in early-stage CC patients prior to radical hysterectomy (RH) with bilateral pelvic lymphadenectomy (BPL), in which positive lymph node metastasis decreasing overall survival (OS) from 80% to 53% at 5 years.

MicroRNAs (miRNAs) are single-strand RNAs comprising approximately 21-23 nucleotides. miRNAs regulate gene expression through the inhibition of posttranscriptional events and, in some cases, induce the degradation of their target messenger RNA. In cancer, miRNAs can function as both oncogenes and/or as tumor suppressor genes depending on the function of their target genes.

Formalin-fixed paraffin-embedded (FFPE) tissue blocks from CC patients diagnosed between January 2006 and December 2013 at the Department of Oncologic Gynecology of the National Cancer Institute (Mexico City) were analyzed with the intention of selecting those with a confirmed histopathological diagnosis of stages IB1 or IIA1 CC treated with RH and BPL. Total RNA was extracted from 5 (10-µm) sections for selected tissues.For the clinical correlation analysis, the samples were divided into 2 groups: 1 with positive occult lymph node metastasis pathology and 1 without lymph node metastasis pathology. For both groups, patients were matched for age, tumor size and presence of lymphovascular permeation.

The identification of global miRNA profiles was performed using GeneChip miRNA 3.0 Array (Affymetrix, Cat. 902018) following the manufacturer's instructions. the microarray was hybridized and washed using the Affymetrix Fluidics Station 450 and scanned with the Affymetrix GeneChip Scanner 3000. After processing the images, the raw data were processed. To obtain the miRNA profile, the processed samples were divided into 2 groups, samples with lymph node metastasis and samples without lymph node metastasis. Differentially expressed miRNAs were identified using a cutoff value of p <0.01 and a fold change (FC) of 1.5. miRNAs that met these criteria were classified as over-expressed or under-expressed.

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer histopathological diagnosis
* Clinical stage IB1 or IIA1 CC
* Treated with radical hysterectomy (RH) with bilateral pelvic lymphadenectomy (BPL)

Exclusion Criteria:

* Double primary tumors
* Treatment regimens other than standard treatment
* Poor quality formalin-fixed paraffin-embedded tissue blocks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cervical cancer between January 2006 and December 2013 at the Department of Oncologic Gynecology of the National Cancer Institute (Mexico City).
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Prognostic miRNAs | 7 years
  Identify a subset of miRNAs with prognostic value associated with early-stage CC patients treated with RH and BPL with positive lymph node metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: David F Cantú-deLeón, MD, PhD, Principal Investigator — National Cancer Institute of Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomison J 3rd, Thomas LK, Shroyer KR. Human papillomavirus: molecular and cytologic/histologic aspects related to cervical intraepithelial neoplasia and carcinoma. Hum Pathol. 2008 Feb;39(2):154-66. doi: 10.1016/j.humpath.2007.11.002. PMID 18206494
- [Background] Koh WJ, Greer BE, Abu-Rustum NR, Apte SM, Campos SM, Chan J, Cho KR, Cohn D, Crispens MA, DuPont N, Eifel PJ, Gaffney DK, Giuntoli RL 2nd, Han E, Huh WK, Lurain JR 3rd, Martin L, Morgan MA, Mutch D, Remmenga SW, Reynolds RK, Small W Jr, Teng N, Tillmanns T, Valea FA, McMillian NR, Hughes M; National Comprehensive Cancer Network. Cervical cancer. J Natl Compr Canc Netw. 2013 Mar 1;11(3):320-43. doi: 10.6004/jnccn.2013.0043. PMID 23486458
- [Background] Lea JS, Lin KY. Cervical cancer. Obstet Gynecol Clin North Am. 2012 Jun;39(2):233-53. doi: 10.1016/j.ogc.2012.02.008. Epub 2012 Apr 24. PMID 22640713
- [Background] Delgado G, Bundy B, Zaino R, Sevin BU, Creasman WT, Major F. Prospective surgical-pathological study of disease-free interval in patients with stage IB squamous cell carcinoma of the cervix: a Gynecologic Oncology Group study. Gynecol Oncol. 1990 Sep;38(3):352-7. doi: 10.1016/0090-8258(90)90072-s. PMID 2227547
- [Background] Suprasert P, Charoenkwan K, Khunamornpong S. Pelvic node removal and disease-free survival in cervical cancer patients treated with radical hysterectomy and pelvic lymphadenectomy. Int J Gynaecol Obstet. 2012 Jan;116(1):43-6. doi: 10.1016/j.ijgo.2011.08.001. Epub 2011 Oct 5. PMID 21978816
- [Background] Togami S, Kamio M, Yanazume S, Yoshinaga M, Douchi T. Can pelvic lymphadenectomy be omitted in stage IA2 to IIB uterine cervical cancer? Int J Gynecol Cancer. 2014 Jul;24(6):1072-6. doi: 10.1097/IGC.0000000000000163. PMID 24905616
- [Background] Tanaka Y, Sawada S, Murata T. Relationship between lymph node metastases and prognosis in patients irradiated postoperatively for carcinoma of the uterine cervix. Acta Radiol Oncol. 1984;23(6):455-9. doi: 10.3109/02841868409136048. PMID 6099039
- [Background] Bartel DP. MicroRNAs: genomics, biogenesis, mechanism, and function. Cell. 2004 Jan 23;116(2):281-97. doi: 10.1016/s0092-8674(04)00045-5. PMID 14744438
- [Background] Pedroza-Torres A, Lopez-Urrutia E, Garcia-Castillo V, Jacobo-Herrera N, Herrera LA, Peralta-Zaragoza O, Lopez-Camarillo C, De Leon DC, Fernandez-Retana J, Cerna-Cortes JF, Perez-Plasencia C. MicroRNAs in cervical cancer: evidences for a miRNA profile deregulated by HPV and its impact on radio-resistance. Molecules. 2014 May 16;19(5):6263-81. doi: 10.3390/molecules19056263. PMID 24840898
- [Background] Lee JW, Choi CH, Choi JJ, Park YA, Kim SJ, Hwang SY, Kim WY, Kim TJ, Lee JH, Kim BG, Bae DS. Altered MicroRNA expression in cervical carcinomas. Clin Cancer Res. 2008 May 1;14(9):2535-42. doi: 10.1158/1078-0432.CCR-07-1231. PMID 18451214
- See also: GLOBOCAN 2012 v1.0, Cancer Incidence and Mortality Worldwide: IARC CancerBase. No. 11 [Internet]., Lyon, Fr. Int. Agency Res. Cancer. 11 (2013) — http://gco.iarc.fr